CLINICAL TRIAL: NCT00552474
Title: A Clinical Evaluation of Bilateral Stimulation of the Subthalamic Nucleus (STN) Using the ANS Totally Implantable Deep Brain Stimulation System as an Adjunctive Treatment for Reducing Some of the Symptoms of Advanced, Levodopa-responsive Parkinson's Disease That Are Not Adequately Controlled With Medication.
Brief Title: Deep Brain Stimulation to Treat Symptoms of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-04-01
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease; Movement Disorders
Keywords: Parkinson disease; Movement disorders; Deep Brain Stimulation; Libra; l-dopa; levodopa; neuromodulation; neurostimulation; Electrical stimulation of the brain; STN; Subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Placebo Comparator): Implanted but no active stimulation
  Interventions: Device: Libra Deep Brain Stimulation System
- Group A (Experimental): Active Stimulation
  Interventions: Device: Libra Deep Brain Stimulation System

INTERVENTIONS:
Device: Libra Deep Brain Stimulation System — Active DBS Therapy
  Arms: Group A
Device: Libra Deep Brain Stimulation System — Implanted system but no stimulation
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of bilateral stimulation of the subthalamic nucleus (STN) of the brain when using the ANS Totally Implantable Deep Brain Stimulation System as an adjunctive treatment for reducing some of the symptoms of Parkinson's Disease that are not adequately controlled with medication.

DETAILED DESCRIPTION:
This is a prospective, controlled, multi-centered, 12 months post-implantation study. A maximum of 15 sites will enroll a total of 136 patients.

All study participants will have the study device surgically implanted. After implant surgery, study participants will return to the clinic for evaluation 30 days after surgery, three months after surgery, six months after surgery and twelve months after surgery. At the baseline, three, six and twelve month visits the patient's Parkinson's symptoms and ability to perform daily activities will be evaluated using a number of accepted assessment tools including a Dyskinesia diary, evaluation of PD symptoms, quality of life scoring and patient extension study to monitor the safety and efficacy of the ANS Libra/Libra Deep Brain Stimulation System.

After the 1 year study, patients may enter another protocol (C-06-04) to continue to monitor the safety and efficacy of the Libra Deep Brain Stimulation System. Patients may be followed for an additional 4 years.

If necessary, patients may continue to have access to the investigational device under protocol (C-13-02) which allows for compassionate use access to it.

ELIGIBILITY:
Inclusion Criteria:

* Person is 18 to 80 years of age
* Person has been diagnosed with Parkinson's disease for at lease five (5) years
* Person experiences at least six (6) hours or more daily "off-time" or moderate to severe dyskinesias during waking hours
* Person has a history of improvement of Parkinson's symptoms with l-dopa (levodopa) therapy
* Person must be willing to maintain a constant dose of anti-Parkinson's disease medication for at least one month prior to study enrollment
* Person must be available for appropriate follow-up times for the length of the study

Exclusion Criteria:

* Person has any major illness or medical condition that would interfere with participation in the study
* Person currently suffers from untreated, major depression
* Person has an electrical or electromagnetic implant (e.g. cochlear prosthesis or pacemaker)
* Person has had a prior surgery for the treatment of PD symptoms, including previous DBS surgery
* Person has dementia
* Person has a history of seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Increase the duration of "on time" without dyskinesias or with non-bothersome dyskinesias | 90 days

SECONDARY OUTCOMES:
Changes in the following over time: Incidence of AEs; UPDRS motor scores; Activities of Daily Living; Quality of Life, Quality Sleep Index, Hoehn and Yahr Staging, Global Outcome evaluation and Patient Satisfaction | 1 year

OTHER OUTCOMES:
Efficacy | Yearly for 5 years
  Reduction in Parkinson's symptoms as demonstrated by the total UPDRS scores and each individual component of the UPDRS in the medication on and off state with stimulation on at 2 years, 3 years, 4 years, and 5 years.
Quality of life | up to to 5 years
  Quality of Life measurements as measured by the Parkinson's Disease Questionnaire (PDQ 39)
Activites of Daily Living | up to 5 years
  Activities of Daily Living measurement at 2 years, 3 years, 4 years, and 5 years as determined from the Unified Parkinson's Disease Rating Scale (UPDRS) in the medication on and stimulation on state

CONTACTS AND LOCATIONS:
Overall Officials: DeLea Peichel, Study Director — ANS/St Jude Medical
Locations (15):
- United States (15):
  - Loma Linda University School of Medicine, Loma Linda, California
  - University of Florida, Gainesville, Florida
  - Universtiy of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Lahey Clinic, Burlington, Massachusetts
  - Oakwood Hospital, Dearborn, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Mayfield Clinic, Cincinnati, Ohio
  - Pennsylvania Hospital (UPHS), Philadelphia, Pennsylvania
  - Neurology Specialists of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Univerisity of Virginia, Charlottesville, Virginia
  - Medical College of Wisconcin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Okun MS, Gallo BV, Mandybur G, Jagid J, Foote KD, Revilla FJ, Alterman R, Jankovic J, Simpson R, Junn F, Verhagen L, Arle JE, Ford B, Goodman RR, Stewart RM, Horn S, Baltuch GH, Kopell BH, Marshall F, Peichel D, Pahwa R, Lyons KE, Troster AI, Vitek JL, Tagliati M; SJM DBS Study Group. Subthalamic deep brain stimulation with a constant-current device in Parkinson's disease: an open-label randomised controlled trial. Lancet Neurol. 2012 Feb;11(2):140-9. doi: 10.1016/S1474-4422(11)70308-8. Epub 2012 Jan 11. PMID 22239915
- See also: ANS specific website — http://www.ans-medical.com